CLINICAL TRIAL: NCT02171052
Title: Relative Bioavailability of Dabigatran and Digoxin After 150 mg BID Dabigatran Etexilate and Digoxin at 0.25 mg QD Alone or Following Concomitant Multiple Oral Administrations in Healthy Male and Female Volunteers (an Open Label, Randomised, Multiple-dose, Three-way Crossover Study)
Brief Title: Relative Bioavailability of Dabigatran and Digoxin in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.59
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Digoxin

ARMS (3):
- Dabigatran etexilate plus digoxin (Experimental)
  Interventions: Drug: Dabigatran etexilate; Drug: Digoxin
- Dabigatran etexilate (Active Comparator)
  Interventions: Drug: Dabigatran etexilate
- Digoxin (Active Comparator)
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Dabigatran etexilate
  Arms: Dabigatran etexilate; Dabigatran etexilate plus digoxin
Drug: Digoxin
  Arms: Dabigatran etexilate plus digoxin; Digoxin

SUMMARY:
To investigate the bioavailability of dabigatran with and without concomitant administration of digoxin and the bioavailability of digoxin with and without concomitant administration of dabigatran etexilate

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and ≤65 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder or acute blood coagulation defect
4. Puls below 50 bpm at screening
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
9. Intake of any medication within four weeks of first dosing.
10. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within four weeks prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Within 5 days of study medication no intake of grapefruit, grapefruit juice, or products containing grapefruit juice, Seville oranges, garlic supplements, or St. John's Worth
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. Excessive physical activities (within one week prior to administration or during the trial)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. Females of child bearing potential who are pregnant, breast feeding or who are either not surgically sterile or are sexually active and not using an acceptable form of contraception as either the oral contraceptives since at least two months and the double barrier method, i.e. intrauterine device with spermicide and condom for the male partner
20. Male subjects must agree to minimise the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the post study medical. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)
21. Planned surgeries within four weeks following the end-of study examination
22. Intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, cumarin etc.
23. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
24. Vulnerable subjects (e.g. persons kept in detention).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to 72 hours after drug administration on day 4
Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) | 2 hours before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after drug administration on day 4

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma from the time point 0 after the last dose at steady state to the last quantifiable analyte plasma concentration within the uniform dosing interval τ (AUC0-tz,ss) | Up to 72 hours after drug administration on day 4
Time of last measurable concentration of the analyte in plasma within the dosing interval τ at steady state (tz,ss) | Up to 72 hours after drug administration on day 4
Time from last dosing to the maximum concentration of the analyte in plasma at steady state (tmax,ss) | Up to 72 hours after drug administration on day 4
Apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration (CL/Fss) | Up to 72 hours after drug administration on day 4
Renal clearance of the analyte at steady state determined over the dosing interval τ (CLR,ss) | Up to 24 hours after drug administration on day 4
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Up to 72 hours after drug administration on day 4
Time from last dosing to the minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ ( tmin,ss) | Up to 72 hours after drug administration on day 4
Pre-dose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) | 2 hours before drug administration on day 4
Mean residence time of the analyte in the body at steady state after p.o. administration (MRTp.o.,ss) | Up to 72 hours after drug administration on day 4
Fraction of parent drug eliminated in urine at steady state over a uniform dosing interval τ (feτ,ss) | Up to 24 hours after drug administration on day 4
Assessment of tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | Day 76
Apparent volume of distribution during the terminal phase λz at steady state following an extravascular administration (Vz/Fss) | Up to day 7
Amount of analyte that was eliminated in urine at steady state over an uniform dosing interval τ (Aeτ,ss) | Up to 24 hours after drug administration on day 4
Area under the effect ratio curve (AUERτ,ss) for activated prothrombin time (aPTT) and ecarin clotting time (ECT) | Up to 72 hours after drug administration on day 4
Prolongation at trough (ERpre,ss) for aPTT | Up to 72 hours after drug administration on day 4
Change from baseline in physical examination | Baseline, day 76
Change from baseline in vital signs (blood pressure, pulse rate) | Baseline, day 76
Change from baseline in 12-lead electrocardiogram | Baseline, day 76
Change from baseline in clinical laboratory tests | Baseline, day 76
Number of Participants with Serious and Non-Serious Adverse Events | Up to day 76
Maximum effect ratio at steady state (ERmax,ss) for aPTT and ECT | Up to 72 hours after drug administration on day 4
Prolongation at trough (ERpre,ss) for ECT | Up to 72 hours after drug administration on day 4